CLINICAL TRIAL: NCT03084718
Title: An 8-week, Multicenter, Randomized, Double-blind, Placebo and Active-controlled, Parallel Group, Dose-ranging Study to Evaluate the Efficacy and Safety of 3 Doses of CHF 718 pMDI (HFA Beclomethasone Dipropionate Via Pressured Metered Dose Inhaler) in Asthmatic Subjects.
Brief Title: An 8-week Dose Ranging Study of CHF 718 pMDI in Asthmatic Subjects
Acronym: BEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CCD-05993AA3-01
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A (Experimental): CHF 718 pMDI 100 μg Total Daily Dose (TDD), Dose 1; CHF 718 pMDI 50 μg/actuation: 1 inhalation twice daily (BID);
  Interventions: Drug: CHF 718 pMDI
- Treatment B (Experimental): CHF 718 pMDI 400 μg Total Daily Dose (TDD) 400 μg, Dose 2; CHF 718 pMDI 100 μg/actuation: 2 inhalations BID;
  Interventions: Drug: CHF 718 pMDI
- Treatment C (Experimental): CHF 718 pMDI Total Daily Dose (TDD) 800 μg, Dose 3; CHF 718 pMDI 100 μg/actuation: 4 inhalations BID;
  Interventions: Drug: CHF 718 pMDI
- Treatment D (Placebo Comparator): Placebo Control, Placebo; CHF 718 pMDI matched Placebo: 4 inhalations BID;
  Interventions: Drug: Placebo pMDI
- Treatment E (Active Comparator): Beclomethasone dipropionate (BDP) Hydrofluoroalkane (HFA), Total Daily Dose (TDD) 320 µg; QVAR® 80 μg/actuation: 2 inhalations BID;
  Interventions: Drug: Beclomethasone Dipropionate (BDP)

INTERVENTIONS:
Drug: CHF 718 pMDI — Dose Response: Test one of three different doses of CHF 718 pMDI
  Arms: Treatment A; Treatment B; Treatment C
Drug: Placebo pMDI — Placebo Control
  Arms: Treatment D
Drug: Beclomethasone Dipropionate (BDP) — Active Control
  Other Names: QVAR® 80µg
  Arms: Treatment E

SUMMARY:
The purpose of this study is to evaluate the dose-response of different doses of CHF 781 Pressurized Metered Dose Inhaler (pMDI) on lung function and other clinical outcomes, to identify the optimal dose(s) in terms of benefit/ risk ratio for further development in the target patient population.

DETAILED DESCRIPTION:
This is a phase II, multicenter, randomized, double-blind, placebo and active controlled dose ranging 5-arm parallel group study to identify the optimal dose of CHF 781 pMDI with respect to lung function and other clinical efficacy and safety outcomes.

After a 2 week run-in period under rescue albuterol as needed and background inhaled corticosteroid (ICS), patients will be randomized to one of the 5 study treatment groups. After randomization, patients will be assessed after 4 and 8 weeks of study treatment at the center. A follow-up phone call will be performed a week after the last visit.

During the study, daily asthma symptoms, peak expiratory flow, rescue and background medication use, and compliance with the study medication will be recorded via subject diary. Treatment-Emergent Adverse Events (TEAEs) will be assessed and recorded throughout the study. At screening and subsequent visits, patients will undergo physical and vital signs examinations, spirometry measurements, and 12-lead ECG. Routine hematology, blood chemistry, and pregnancy testing will be performed before enrollment and at end of study. 24-hr urine cortisol and creatinine will be assessed before and after the first dose and just before the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 and ≤75 years who have signed an Informed Consent form prior to initiation of any study-related procedure.
* A diagnosis of asthma as defined in the Global Initiative for Asthma (GINA) Report, 2016, documented for at least 1 year prior to screening.
* Subjects with poorly controlled or uncontrolled asthma evidenced by a score at the Asthma Control Questionnaire 7 © (ACQ-7) ≥1.5 (this criterion must be met at screening and at randomization visits).
* Subjects with a pre-bronchodilator Forced Expiratory Volume in the 1st Second (FEV1) ≥50% and <85% of their predicted normal value, after appropriate washout from bronchodilators, at the screening and randomization visits.
* Subjects with a positive response to a reversibility test at screening (pre - post BD), within 1 year prior to or at screening defined as ΔFEV1≥12% and ≥200 mL over baseline within 30 minutes after inhaling 4 puffs of albuterol HFA 90µg/actuation.
* Use of inhaled corticosteroids (low/medium dose according to GINA Report 2016) with or without a long-acting bronchodilator (LABD) for 3 months (stable dose in the last 4 weeks) before screening visit (V).
* A cooperative attitude and ability to demonstrate correct use of the diary, peak flow meter, and pMDI inhalers.
* A basal morning (7-10 am) serum cortisol level between 7-28 µg/dL at screening visit (V1).
* A Body Mass Index (BMI): 18.5 ≤ BMI <35 kg/m^2.

Exclusion Criteria:

* Pregnant (as evident by a positive urine human chorionic gonadotropin (hCG) or serum β-hCG test) or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they are willing to use a highly effective birth control method
* Subjects who suffer from chronic obstructive pulmonary disease (COPD) as defined by the GOLD Report 2017, or are suspected of having Asthma COPD Overlap Syndrome (ACOS) as defined in GINA Report, 2016.
* Inability to carry out pulmonary lung function testing, to comply with study procedures or with study drug intake.
* Current smokers or ex-smokers (tobacco, vapor cigarettes, marijuana) with a smoking history of >10 pack-years or having stopped smoking one year or less prior to screening visit.
* History of life-threatening asthma, clinically significant uncontrolled disease or respiratory infection.
* An asthma exacerbation requiring oral corticosteroids within 3 months or hospitalization within 6 months prior to screening.
* Subjects with unresolved bacterial or viral respiratory tract, sinus or middle ear infection affecting asthma status within 2 weeks prior to screening.
* Subjects who received a vaccination within 2 weeks prior to screening or during the run-in.
* Subjects with oral candidiasis at screening or at randomization.
* Subjects with any clinically significant, uncontrolled condition
* Subjects who have clinically significant cardiovascular condition
* Subjects who have a clinically significant abnormal 12-lead ECG that results in active medical problem which may impact the safety of the subject according to Investigator's judgement.
* Subjects whose 12-lead ECG shows Fridericia corrected QT interval (QTcF) >450 ms for males or QTcF >470 ms for females at screening and randomization visits.
* Subjects with known intolerance/hypersensitivity or contra-indication to treatment with ß2-adrenergic receptor agonists, inhaled corticosteroids or propellant gases/excipients.
* Subjects with concomitant immunosuppressive therapy, use of oral or injected corticosteroids, anti-Immunoglobulin E (IgE), anti-Interleukin 5 (IL5), or other monoclonal or polyclonal antibodies within 12 weeks prior to screening.
* Use of potent cytochrome P450 3A4 inhibitors and inducers within 4 weeks prior to screening.
* History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening.
* Subjects who have received an investigational drug within 1 month or 5 half-lives (whichever is greater) prior to screening visit, or have been previously randomized in this trial, or are currently participating in another clinical trial.
* Subjects who are mentally or legally incapacitated, or subjects accommodated in an establishment as a result of an official or judicial order.
* Subjects who have undergone major surgery in the 3 months prior to screening visit or have a planned surgery during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bernstein, MD, Principal Investigator — Bernstein Clinical Research Center, LLC
Locations (114):
- United States (114):
  - Chiesi Investigational Site, Birmingham, Alabama
  - Chiesi Investigational Site, Montgomery, Alabama
  - Chiesi Investigational Site, Phoenix, Arizona
  - Chiesi Investigational Site, Surprise, Arizona
  - Chiesi Investigational Site, Tempe, Arizona
  - Chiesi Investigational Site, Little Rock, Arkansas
  - Chiesi Investigational Site, Anaheim, California
  - Chiesi Investigational Site, Encinitas, California
  - Chiesi Investigational Site, Escondido, California
  - Chiesi Investigational Site, Fullerton, California
  - Chiesi Investigational Site, Huntington Beach, California
  - Chiesi Investigational Site, Long Beach, California
  - Chiesi Investigational Site, Los Angeles, California
  - Chiesi Investigational Site, Newport Beach, California
  - Chiesi Investigational Site, North Hollywood, California
  - Chiesi Investigational Site, Rolling Hills Estates, California
  - Chiesi Investigational Site, Sacramento, California
  - Chiesi Investigational Site, San Diego, California
  - Chiesi Investigational Site, San Jose, California
  - Chiesi Investigational Site, Tustin, California
  - Chiesi Investigational Site, Westminster, California
  - Chiesi Investigational Site, Boulder, Colorado
  - Chiesi Investigational Site, Colorado Springs, Colorado
  - Chiesi Investigational Site, Denver, Colorado
  - Chiesi Investigational Site, Greenwood, Colorado
  - Chiesi Investigational Site, Wheat Ridge, Colorado
  - Chiesi Investigational Site, Aventura, Florida
  - Chiesi Investigational Site, Clearwater, Florida
  - Chiesi Investigational Site, Daytona Beach, Florida
  - Chiesi Investigational Site, Doral, Florida
  - Chiesi Investigational Site, Gainesville, Florida
  - Chiesi Investigational Site, Hialeah, Florida
  - Chiesi Investigational Site, Kissimmee, Florida
  - Chiesi Investigational Site, Lauderdale Lakes, Florida
  - Chiesi Investigational Site, Loxahatchee Groves, Florida
  - Chiesi Investigational Site, Maitland, Florida
  - Chiesi Investigational Site, Miami, Florida
  - Chiesi Investigational Site, Orlando, Florida
  - Chiesi Investigational Site, Palmetto Bay, Florida
  - Chiesi Investigational Site, Plantation, Florida
  - Chiesi Investigational Site, Pompano Beach, Florida
  - Chiesi Investigational Site, Saint Cloud, Florida
  - Chiesi Investigational Site, Sarasota, Florida
  - Chiesi Investigational Site, Winter Park, Florida
  - Chiesi Investigational Site, Dacula, Georgia
  - Chiesi Investigational Site, Duluth, Georgia
  - Chiesi Investigational Site, Gainesville, Georgia
  - Chiesi Investigational Site, Marietta, Georgia
  - Chiesi Investigational Site, Savannah, Georgia
  - Chiesi Investigational Site, Chicago, Illinois
  - Chiesi Investigational Site, Crowley, Louisiana
  - Chiesi Investigational Site, New Orleans, Louisiana
  - Chiesi Investigational Site, Baltimore, Maryland
  - Chiesi Investigational Site, Bethesda, Maryland
  - Chiesi Investigational Site, Fall River, Massachusetts
  - Chiesi Investigational Site, North Dartmouth, Massachusetts
  - Chiesi Investigational Site, South Dartmouth, Massachusetts
  - Chiesi Investigational Site, Detroit, Michigan
  - Chiesi Investigational Site, Minneapolis, Minnesota
  - Chiesi Investigational Site, Columbia, Missouri
  - Chiesi Investigational Site, Festus, Missouri
  - Chiesi Investigational Site, Rolla, Missouri
  - Chiesi Investigational Site, St Louis, Missouri
  - Chiesi Investigational Site, Warrensburg, Missouri
  - Chiesi Investigational Site, Missoula, Montana
  - Chiesi Investigational Site, Omaha, Nebraska
  - Chiesi Investigational Site, Las Vegas, Nevada
  - Chiesi Investigational Site, Skillman, New Jersey
  - Chiesi Investigational Site, Albuquerque, New Mexico
  - Chiesi Investigational Site, Brooklyn, New York
  - Chiesi Investigational Site, New York, New York
  - Chiesi Investigational Site, The Bronx, New York
  - Chiesi Investigational Site, Charlotte, North Carolina
  - Chiesi Investigational Site, Gastonia, North Carolina
  - Chiesi Investigational Site, Hendersonville, North Carolina
  - Chiesi Investigational Site, Hickory, North Carolina
  - Chiesi Investigational Site, Monroe, North Carolina
  - Chiesi Investigational Site, Mooresville, North Carolina
  - Chiesi Investigational Site, Winston-Salem, North Carolina
  - Chiesi Investigational Site, Cincinnati, Ohio
  - Chiesi Investigational Site, Dayton, Ohio
  - Chiesi Investigational Site, Grove City, Ohio
  - Chiesi Investigational Site, Munroe Falls, Ohio
  - Chiesi Investigational Site, Toledo, Ohio
  - Chiesi Investigational Site, Edmond, Oklahoma
  - Chiesi Investigational Site, Medford, Oregon
  - Chiesi Investigational Site, Portland, Oregon
  - Chiesi Investigational Site, East Providence, Rhode Island
  - Chiesi Investigational Site, Warwick, Rhode Island
  - Chiesi Investigational Site, Anderson, South Carolina
  - Chiesi Investigational Site, Gaffney, South Carolina
  - Chiesi Investigational Site, Greenville, South Carolina
  - Chiesi Investigational Site, Rock Hill, South Carolina
  - Chiesi Investigational Site, Spartanburg, South Carolina
  - Chiesi Investigational Site, Union, South Carolina
  - Chiesi Investigational Site, Chattanooga, Tennessee
  - Chiesi Investigational Site, Knoxville, Tennessee
  - Chiesi Investigational Site, Smyrna, Tennessee
  - Chiesi Investigational Site, Spring Hill, Tennessee
  - Chiesi Investigational Site, Allen, Texas
  - Chiesi Investigational Site, Beaumont, Texas
  - Chiesi Investigational Site, Cypress, Texas
  - Chiesi Investigational Site, Dallas, Texas
  - Chiesi Investigational Site, El Paso, Texas
  - Chiesi Investigational Site, McKinney, Texas
  - Chiesi Investigational Site, Pearland, Texas
  - Chiesi Investigational Site, Plano, Texas
  - Chiesi Investigational Site, San Antonio, Texas
  - Chiesi Investigational Site, Sherman, Texas
  - Chiesi Investigational Site, St. George, Utah
  - Chiesi Investigational Site, South Burlington, Vermont
  - Chiesi Investigational Site, Norfolk, Virginia
  - Chiesi Investigational Site, Everett, Washington
  - Chiesi Investigational Site, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tilert T, Dillon C, Paulose-Ram R, Hnizdo E, Doney B. Estimating the U.S. prevalence of chronic obstructive pulmonary disease using pre- and post-bronchodilator spirometry: the National Health and Nutrition Examination Survey (NHANES) 2007-2010. Respir Res. 2013 Oct 9;14(1):103. doi: 10.1186/1465-9921-14-103. PMID 24107140
- [Background] Mannino DM. COPD: epidemiology, prevalence, morbidity and mortality, and disease heterogeneity. Chest. 2002 May;121(5 Suppl):121S-126S. doi: 10.1378/chest.121.5_suppl.121s. PMID 12010839
- [Background] Tonnesen P. Smoking cessation and COPD. Eur Respir Rev. 2013 Mar 1;22(127):37-43. doi: 10.1183/09059180.00007212. PMID 23457163
- [Background] van Eerd EA, van der Meer RM, van Schayck OC, Kotz D. Smoking cessation for people with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2016 Aug 20;2016(8):CD010744. doi: 10.1002/14651858.CD010744.pub2. PMID 27545342
- [Background] Kew KM, Mavergames C, Walters JA. Long-acting beta2-agonists for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2013 Oct 15;2013(10):CD010177. doi: 10.1002/14651858.CD010177.pub2. PMID 24127118
- [Background] McGarvey L, Niewoehner D, Magder S, Sachs P, Tetzlaff K, Hamilton A, Korducki L, Bothner U, Vogelmeier C, Koch A, Ferguson GT. One-Year Safety of Olodaterol Once Daily via Respimat(R) in Patients with GOLD 2-4 Chronic Obstructive Pulmonary Disease: Results of a Pre-Specified Pooled Analysis. COPD. 2015;12(5):484-93. doi: 10.3109/15412555.2014.991864. Epub 2015 Feb 18. PMID 25692310
- [Background] Dahl R, Chung KF, Buhl R, Magnussen H, Nonikov V, Jack D, Bleasdale P, Owen R, Higgins M, Kramer B; INVOLVE (INdacaterol: Value in COPD: Longer Term Validation of Efficacy and Safety) Study Investigators. Efficacy of a new once-daily long-acting inhaled beta2-agonist indacaterol versus twice-daily formoterol in COPD. Thorax. 2010 Jun;65(6):473-9. doi: 10.1136/thx.2009.125435. PMID 20522841
- [Background] Keating GM. Tiotropium bromide inhalation powder: a review of its use in the management of chronic obstructive pulmonary disease. Drugs. 2012 Jan 22;72(2):273-300. doi: 10.2165/11208620-000000000-00000. PMID 22217233
- [Background] Casaburi R, Kukafka D, Cooper CB, Witek TJ Jr, Kesten S. Improvement in exercise tolerance with the combination of tiotropium and pulmonary rehabilitation in patients with COPD. Chest. 2005 Mar;127(3):809-17. doi: 10.1378/chest.127.3.809. PMID 15764761
- [Background] Kesten S, Casaburi R, Kukafka D, Cooper CB. Improvement in self-reported exercise participation with the combination of tiotropium and rehabilitative exercise training in COPD patients. Int J Chron Obstruct Pulmon Dis. 2008;3(1):127-36. doi: 10.2147/copd.s2389. PMID 18488436
- [Background] Karner C, Chong J, Poole P. Tiotropium versus placebo for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009285. doi: 10.1002/14651858.CD009285.pub2. PMID 22786525
- [Background] Wedzicha JA, Banerji D, Chapman KR, Vestbo J, Roche N, Ayers RT, Thach C, Fogel R, Patalano F, Vogelmeier CF; FLAME Investigators. Indacaterol-Glycopyrronium versus Salmeterol-Fluticasone for COPD. N Engl J Med. 2016 Jun 9;374(23):2222-34. doi: 10.1056/NEJMoa1516385. Epub 2016 May 15. PMID 27181606
- [Background] Yang IA, Clarke MS, Sim EH, Fong KM. Inhaled corticosteroids for stable chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD002991. doi: 10.1002/14651858.CD002991.pub3. PMID 22786484
- [Background] Pavord ID, Lettis S, Locantore N, Pascoe S, Jones PW, Wedzicha JA, Barnes NC. Blood eosinophils and inhaled corticosteroid/long-acting beta-2 agonist efficacy in COPD. Thorax. 2016 Feb;71(2):118-25. doi: 10.1136/thoraxjnl-2015-207021. Epub 2015 Nov 19. PMID 26585525
- [Background] Kew KM, Seniukovich A. Inhaled steroids and risk of pneumonia for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2014 Mar 10;2014(3):CD010115. doi: 10.1002/14651858.CD010115.pub2. PMID 24615270
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Yawn BP, Li Y, Tian H, Zhang J, Arcona S, Kahler KH. Inhaled corticosteroid use in patients with chronic obstructive pulmonary disease and the risk of pneumonia: a retrospective claims data analysis. Int J Chron Obstruct Pulmon Dis. 2013;8:295-304. doi: 10.2147/COPD.S42366. Epub 2013 Jun 27. PMID 23836970
- [Background] Rachelefsky GS, Liao Y, Faruqi R. Impact of inhaled corticosteroid-induced oropharyngeal adverse events: results from a meta-analysis. Ann Allergy Asthma Immunol. 2007 Mar;98(3):225-38. doi: 10.1016/S1081-1206(10)60711-9. PMID 17378253
- [Background] Roland NJ, Bhalla RK, Earis J. The local side effects of inhaled corticosteroids: current understanding and review of the literature. Chest. 2004 Jul;126(1):213-9. doi: 10.1378/chest.126.1.213. PMID 15249465
- [Background] Tashkin DP, Murray HE, Skeans M, Murray RP. Skin manifestations of inhaled corticosteroids in COPD patients: results from Lung Health Study II. Chest. 2004 Oct;126(4):1123-33. doi: 10.1016/S0012-3692(15)31287-3. PMID 15486373
- [Background] Crim C, Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Willits LR, Yates JC, Vestbo J. Pneumonia risk in COPD patients receiving inhaled corticosteroids alone or in combination: TORCH study results. Eur Respir J. 2009 Sep;34(3):641-7. doi: 10.1183/09031936.00193908. Epub 2009 May 14. PMID 19443528
- [Background] Crim C, Dransfield MT, Bourbeau J, Jones PW, Hanania NA, Mahler DA, Vestbo J, Wachtel A, Martinez FJ, Barnhart F, Lettis S, Calverley PM. Pneumonia risk with inhaled fluticasone furoate and vilanterol compared with vilanterol alone in patients with COPD. Ann Am Thorac Soc. 2015 Jan;12(1):27-34. doi: 10.1513/AnnalsATS.201409-413OC. PMID 25490706
- [Background] Pavord ID, Lettis S, Anzueto A, Barnes N. Blood eosinophil count and pneumonia risk in patients with chronic obstructive pulmonary disease: a patient-level meta-analysis. Lancet Respir Med. 2016 Sep;4(9):731-741. doi: 10.1016/S2213-2600(16)30148-5. Epub 2016 Jul 23. PMID 27460163
- [Background] Johnell O, Pauwels R, Lofdahl CG, Laitinen LA, Postma DS, Pride NB, Ohlsson SV. Bone mineral density in patients with chronic obstructive pulmonary disease treated with budesonide Turbuhaler. Eur Respir J. 2002 Jun;19(6):1058-63. doi: 10.1183/09031936.02.00276602. PMID 12108857
- [Background] Ferguson GT, Calverley PMA, Anderson JA, Jenkins CR, Jones PW, Willits LR, Yates JC, Vestbo J, Celli B. Prevalence and progression of osteoporosis in patients with COPD: results from the TOwards a Revolution in COPD Health study. Chest. 2009 Dec;136(6):1456-1465. doi: 10.1378/chest.08-3016. Epub 2009 Jul 6. PMID 19581353
- [Background] Loke YK, Cavallazzi R, Singh S. Risk of fractures with inhaled corticosteroids in COPD: systematic review and meta-analysis of randomised controlled trials and observational studies. Thorax. 2011 Aug;66(8):699-708. doi: 10.1136/thx.2011.160028. Epub 2011 May 20. PMID 21602540
- [Background] Suissa S, Kezouh A, Ernst P. Inhaled corticosteroids and the risks of diabetes onset and progression. Am J Med. 2010 Nov;123(11):1001-6. doi: 10.1016/j.amjmed.2010.06.019. Epub 2010 Oct 1. PMID 20870201
- [Background] Wang JJ, Rochtchina E, Tan AG, Cumming RG, Leeder SR, Mitchell P. Use of inhaled and oral corticosteroids and the long-term risk of cataract. Ophthalmology. 2009 Apr;116(4):652-7. doi: 10.1016/j.ophtha.2008.12.001. Epub 2009 Feb 25. PMID 19243828
- [Background] Miller DP, Watkins SE, Sampson T, Davis KJ. Long-term use of fluticasone propionate/salmeterol fixed-dose combination and incidence of cataracts and glaucoma among chronic obstructive pulmonary disease patients in the UK General Practice Research Database. Int J Chron Obstruct Pulmon Dis. 2011;6:467-76. doi: 10.2147/COPD.S14247. Epub 2011 Sep 16. PMID 22003292
- [Background] Andrejak C, Nielsen R, Thomsen VO, Duhaut P, Sorensen HT, Thomsen RW. Chronic respiratory disease, inhaled corticosteroids and risk of non-tuberculous mycobacteriosis. Thorax. 2013 Mar;68(3):256-62. doi: 10.1136/thoraxjnl-2012-201772. Epub 2012 Jul 10. PMID 22781123
- [Background] Aaron SD, Vandemheen KL, Fergusson D, Maltais F, Bourbeau J, Goldstein R, Balter M, O'Donnell D, McIvor A, Sharma S, Bishop G, Anthony J, Cowie R, Field S, Hirsch A, Hernandez P, Rivington R, Road J, Hoffstein V, Hodder R, Marciniuk D, McCormack D, Fox G, Cox G, Prins HB, Ford G, Bleskie D, Doucette S, Mayers I, Chapman K, Zamel N, FitzGerald M; Canadian Thoracic Society/Canadian Respiratory Clinical Research Consortium. Tiotropium in combination with placebo, salmeterol, or fluticasone-salmeterol for treatment of chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):545-55. doi: 10.7326/0003-4819-146-8-200704170-00152. Epub 2007 Feb 19. PMID 17310045
- [Background] Singh D, Brooks J, Hagan G, Cahn A, O'Connor BJ. Superiority of "triple" therapy with salmeterol/fluticasone propionate and tiotropium bromide versus individual components in moderate to severe COPD. Thorax. 2008 Jul;63(7):592-8. doi: 10.1136/thx.2007.087213. Epub 2008 Feb 1. PMID 18245142
- [Background] Hanania NA, Crater GD, Morris AN, Emmett AH, O'Dell DM, Niewoehner DE. Benefits of adding fluticasone propionate/salmeterol to tiotropium in moderate to severe COPD. Respir Med. 2012 Jan;106(1):91-101. doi: 10.1016/j.rmed.2011.09.002. Epub 2011 Oct 29. PMID 22040533
- [Background] Frith PA, Thompson PJ, Ratnavadivel R, Chang CL, Bremner P, Day P, Frenzel C, Kurstjens N; Glisten Study Group. Glycopyrronium once-daily significantly improves lung function and health status when combined with salmeterol/fluticasone in patients with COPD: the GLISTEN study, a randomised controlled trial. Thorax. 2015 Jun;70(6):519-27. doi: 10.1136/thoraxjnl-2014-206670. Epub 2015 Apr 3. PMID 25841237
- [Background] Siler TM, Kerwin E, Singletary K, Brooks J, Church A. Efficacy and Safety of Umeclidinium Added to Fluticasone Propionate/Salmeterol in Patients with COPD: Results of Two Randomized, Double-Blind Studies. COPD. 2016;13(1):1-10. doi: 10.3109/15412555.2015.1034256. Epub 2015 Oct 9. PMID 26451734
- [Background] Singh D, Papi A, Corradi M, Pavlisova I, Montagna I, Francisco C, Cohuet G, Vezzoli S, Scuri M, Vestbo J. Single inhaler triple therapy versus inhaled corticosteroid plus long-acting beta2-agonist therapy for chronic obstructive pulmonary disease (TRILOGY): a double-blind, parallel group, randomised controlled trial. Lancet. 2016 Sep 3;388(10048):963-73. doi: 10.1016/S0140-6736(16)31354-X. Epub 2016 Sep 1. PMID 27598678
- [Background] GlaxoSmithKline. Cross Discipline Team Leader Review: Application number 204275Orig1s000; 2013 Apr 1.
- [Background] GlaxoSmithKline. BREO® ELLIPTA® US Prescribing Information. Research Triangle Park, North Carolina; 2015 Apr.
- [Background] Teva Respiratory LLC. QVAR® US Prescribing Information. Horsham, Pennsylvania; 2014 Jul.
- [Background] GlaxoSmithKline. ARNUITY® ELLIPTA® US Prescribing Information. Research Triangle Park, North Carolina; 2014 Aug.
- [Background] Chiesi Farmaceutici S.p.A. A double blind double dummy, multiple dose comparison of two parallel groups comparing a daily dose of extrafine BDP HFA 400µg vs. BDP CFC 1000µg in asthmatic patients over an 8-week treatment period. 2005 Jul;DM/PR/3303/006/03.
- [Background] Busse WW, Brazinsky S, Jacobson K, Stricker W, Schmitt K, Vanden Burgt J, Donnell D, Hannon S, Colice GL. Efficacy response of inhaled beclomethasone dipropionate in asthma is proportional to dose and is improved by formulation with a new propellant. J Allergy Clin Immunol. 1999 Dec;104(6):1215-22. doi: 10.1016/s0091-6749(99)70016-3. PMID 10589004
- [Background] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Woodcock A, Bleecker ER, Busse WW, Lotvall J, Snowise NG, Frith L, Jacques L, Haumann B, Bateman ED. Fluticasone furoate: once-daily evening treatment versus twice-daily treatment in moderate asthma. Respir Res. 2011 Dec 21;12(1):160. doi: 10.1186/1465-9921-12-160. PMID 22188590
- [Background] Anderson WJ, Lipworth BJ. Does body mass index influence responsiveness to inhaled corticosteroids in persistent asthma? Ann Allergy Asthma Immunol. 2012 Apr;108(4):237-42. doi: 10.1016/j.anai.2011.12.006. Epub 2012 Jan 21. PMID 22469442
- [Background] Boulet LP, Franssen E. Influence of obesity on response to fluticasone with or without salmeterol in moderate asthma. Respir Med. 2007 Nov;101(11):2240-7. doi: 10.1016/j.rmed.2007.06.031. Epub 2007 Aug 8. PMID 17686624
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Arievich H, Overend T, Renard D, Gibbs M, Alagappan V, Looby M, Banerji D. A novel model-based approach for dose determination of glycopyrronium bromide in COPD. BMC Pulm Med. 2012 Dec 8;12:74. doi: 10.1186/1471-2466-12-74. PMID 23217058
- [Background] Vanden Burgt JA, Busse WW, Martin RJ, Szefler SJ, Donnell D. Efficacy and safety overview of a new inhaled corticosteroid, QVAR (hydrofluoroalkane-beclomethasone extrafine inhalation aerosol), in asthma. J Allergy Clin Immunol. 2000 Dec;106(6):1209-26. doi: 10.1067/mai.2000.111582. PMID 11112914
- [Background] Aubier M, Wettenger R, Gans SJ. Efficacy of HFA-beclomethasone dipropionate extra-fine aerosol (800 microg day(-1)) versus HFA-fluticasone propionate (1000 microg day(-1)) in patients with asthma. Respir Med. 2001 Mar;95(3):212-20. doi: 10.1053/rmed.2000.1025. PMID 11266239
- [Background] Gross G, Thompson PJ, Chervinsky P, Vanden Burgt J. Hydrofluoroalkane-134a beclomethasone dipropionate, 400 microg, is as effective as chlorofluorocarbon beclomethasone dipropionate, 800 microg, for the treatment of moderate asthma. Chest. 1999 Feb;115(2):343-51. doi: 10.1378/chest.115.2.343. PMID 10027430
- [Background] Matthys H, Nowak D, Hader S, Kunkel G. Efficacy of chlorofluorocarbon-free beclomethasone dipropionate 400 micrograms day-1 delivered as an extrafine aerosol in adults with moderate asthma. Respir Med. 1998 Jun;92 Suppl A:17-22. doi: 10.1016/s0954-6111(98)90213-x. PMID 9850359
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Ellepola AN, Samaranayake LP. Inhalational and topical steroids, and oral candidosis: a mini review. Oral Dis. 2001 Jul;7(4):211-6. PMID 11575870
- [Background] Torres SR, Peixoto CB, Caldas DM, Silva EB, Akiti T, Nucci M, de Uzeda M. Relationship between salivary flow rates and Candida counts in subjects with xerostomia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Feb;93(2):149-54. doi: 10.1067/moe.2002.119738. PMID 11862202
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Hankinson JL, Kawut SM, Shahar E, Smith LJ, Stukovsky KH, Barr RG. Performance of American Thoracic Society-recommended spirometry reference values in a multiethnic sample of adults: the multi-ethnic study of atherosclerosis (MESA) lung study. Chest. 2010 Jan;137(1):138-45. doi: 10.1378/chest.09-0919. Epub 2009 Sep 9. PMID 19741060
- [Background] Hankinson JL, Bang KM. Acceptability and reproducibility criteria of the American Thoracic Society as observed in a sample of the general population. Am Rev Respir Dis. 1991 Mar;143(3):516-21. doi: 10.1164/ajrccm/143.3.516. PMID 2001060
- [Background] Callejas SL, Biddlecombe RA, Jones AE, Joyce KB, Pereira AI, Pleasance S. Determination of the glucocorticoid fluticasone propionate in plasma by automated solid-phase extraction and liquid chromatography-tandem mass spectrometry. J Chromatogr B Biomed Sci Appl. 1998 Nov 6;718(2):243-50. doi: 10.1016/s0378-4347(98)00374-0. PMID 9840434
- [Background] Taylor RL, Machacek D, Singh RJ. Validation of a high-throughput liquid chromatography-tandem mass spectrometry method for urinary cortisol and cortisone. Clin Chem. 2002 Sep;48(9):1511-9. PMID 12194928
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Virchow JC, Backer V, de Blay F, Kuna P, Ljorring C, Prieto JL, Villesen HH. Defining moderate asthma exacerbations in clinical trials based on ATS/ERS joint statement. Respir Med. 2015 May;109(5):547-56. doi: 10.1016/j.rmed.2015.01.012. Epub 2015 Feb 3. PMID 25676887
- [Background] Peters SP, Kunselman SJ, Icitovic N, Moore WC, Pascual R, Ameredes BT, Boushey HA, Calhoun WJ, Castro M, Cherniack RM, Craig T, Denlinger L, Engle LL, DiMango EA, Fahy JV, Israel E, Jarjour N, Kazani SD, Kraft M, Lazarus SC, Lemanske RF Jr, Lugogo N, Martin RJ, Meyers DA, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Chinchilli VM, Bleecker ER; National Heart, Lung, and Blood Institute Asthma Clinical Research Network. Tiotropium bromide step-up therapy for adults with uncontrolled asthma. N Engl J Med. 2010 Oct 28;363(18):1715-26. doi: 10.1056/NEJMoa1008770. Epub 2010 Sep 19. PMID 20979471
- [Background] Mallinckrodt C, Roger J, Chuang-stein C, Molenberghs G, Lane PW, O'Kelly M, et al. Missing data: turning guidance into action. Stat Biopharm Res. 2013;5(4):369-82.
- [Background] Mallinckrodt CH, Kenward MG. Conceptual Considerations regarding Endpoints, Hypotheses, and Analyses for Incomplete Longitudinal Clinical Trial Data. Drug Inf J. 2009; 43(4): 449-58.
- [Background] National Research Council (US) Panel on Handling Missing Data in Clinical Trials. The Prevention and Treatment of Missing Data in Clinical Trials. Washington (DC): National Academies Press (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK209904/ PMID 24983040
- [Background] Leuchs AK, Zinserling J, Brandt A, Wirtz D, Benda N. Choosing Appropriate Estimands in Clinical Trials. Ther Innov Regul Sci. 2015 Jul;49(4):584-592. doi: 10.1177/2168479014567317. PMID 30222440
- [Background] Edwards D, Berry JJ. The efficiency of simulation-based multiple comparisons. Biometrics. 1987 Dec;43(4):913-28. PMID 3427176
- [Result] Montanaro A, Weinstein S, Beaudot C, Scott SM, Georges G. Efficacy and safety of inhaled extrafine beclomethasone dipropionate in adults with asthma: a randomized, parallel-group, dose-ranging study (BEAM). J Asthma. 2022 Jul;59(7):1410-1419. doi: 10.1080/02770903.2021.1928184. Epub 2021 May 24. PMID 34030555
- See also: From the Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2017. — http://goldcopd.org/
- See also: COPD Foundation - What is COPD — http://www.copdfoundation.org/What-is-COPD/Understanding-COPD/What-is-COPD.aspx
- See also: Global Initiative For Asthma - GINA Report 2016 — http://ginasthma.org/wp-content/uploads/2016/04/wms-GINA-2016-main-report-final.pdf
- See also: Centers for Disease Control and Prevention - Most Recent Asthma Data — https://www.cdc.gov/asthma/most_recent_data.htm
- See also: Chiesi Farmaceutici S.p.A. - Respiratory — https://www.chiesi.com/en/air/
- See also: Chiesi Farmaceutici S.p.A - Press Release: Chiesi Farmaceutifici is the first company to submit a marketing authorisation application to the European Medicine Agency for a triple combination for the treatment of COPD — https://www.chiesi.com/en/chiesi-farmaceutici-is-the-first-company-to-submit-a-marketing-authorisation-application-to-the-european-medicine-agency-for-a-triple-combination-for-the-treatment-of-copd-
- See also: Wikipedia entry - Beclomethasone dipropionate — https://en.wikipedia.org/wiki/Beclometasone_dipropionate
- See also: WebMD LLC - Serum Cortisol — http://emedicine.medscape.com/article/2088826-overview
- See also: Quest Diagnostics- Cortisol, Free and Cortisone, 24 Hour Urine with Creatinine — http://www.questdiagnostics.com/testcenter/BUOrderInfo.action?tc=37355&labCode=MET

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A (CHF 718 pMDI 100 µg TDD): CHF 718 pMDI 100 μg Total Daily Dose (TDD), Dose 1;
  CHF 718 pMDI 50 μg/actuation: 1 inhalation twice daily (BID); TDD of BDP: 100 μg;
- Treatment B (CHF 718 pMDI 400 µg TDD): CHF 718 pMDI 400 μg Total Daily Dose (TDD) 400 μg, Dose 2;
  CHF 718 pMDI 100 μg/actuation: 2 inhalations BID; TDD of BDP: 400 μg;
- Treatment C (CHF 718 pMDI 800 µg TDD): CHF 718 pMDI Total Daily Dose (TDD) 800 μg, Dose 3;
  CHF 718 pMDI 100 μg/actuation: 4 inhalations BID; TDD of BDP: 800 μg;
- Treatment D (Placebo): Placebo Control. CHF 718 pMDI matched Placebo: 4 inhalations 2 times a day (BID);
- Treatment E (QVAR^® 320 µg TDD): Beclomethasone dipropionate Hydrofluoroalkane (HFA) (QVAR^®), Active Control
  Beclomethasone dipropionate Hydrofluoroalkane (HFA), Total Daily Dose (TDD) 320 µg; QVAR^® 80 μg/actuation: 2 inhalations BID;
Period: Overall Study
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^® 320 µg TDD)
Started | 120 | 120 | 122 | 124 | 124
Completed | 109 | 110 | 110 | 110 | 120
Not Completed | 11 | 10 | 12 | 14 | 4
Not completed — Withdrawal by Subject | 4 | 3 | 4 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 5 | 5 | 8 | 2
Not completed — Lack of Efficacy | 2 | 0 | 1 | 4 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Randomization error; E-diary non-compliance; Complications with device use | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Demographic characteristics are presented for the Intention-to-treat (ITT) study population; this explains the differences in the randomized patient numbers that are shown in the Participant Flow.
Groups:
- Treatment A: CHF 718 pMDI 100 µg TDD
- Treatment B: CHF 718 pMDI 400 µg TDD
- Treatment C: CHF 718 pMDI 800 µg TDD
- Treatment D: Placebo Control
- Treatment E: Beclomethasone dipropionate Hydrofluoroalkane (HFA) (QVAR^®), Active Control
  Beclomethasone dipropionate Hydrofluoroalkane (HFA), Total Daily Dose (TDD) 320 µg;
  QVAR® 80 μg/actuation: 2 inhalations BID, Total Daily Dose (TDD) of BDP: 320 μg;
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Total
Number analyzed (Participants) | 118 | 116 | 120 | 124 | 124 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 2 | 0 | 2
  Between 18 and 65 years | 97 | 101 | 107 | 110 | 105 | 520
  >=65 years | 21 | 15 | 13 | 12 | 19 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (13.58) | 48.1 (14.38) | 48.2 (13.83) | 45.4 (16.17) | 48.8 (14.24) | 48.1 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 77 | 76 | 72 | 77 | 376
  Male | 44 | 39 | 44 | 52 | 47 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 34 | 30 | 40 | 28 | 166
  Not Hispanic or Latino | 84 | 82 | 90 | 84 | 96 | 436
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 0 | 3
  Asian | 1 | 1 | 0 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 27 | 23 | 28 | 21 | 24 | 123
  White | 78 | 82 | 84 | 93 | 93 | 430
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 7 | 9 | 5 | 41
Region of Enrollment [Number; unit: participants]
  United States | 118 | 116 | 120 | 124 | 124 | 602
Weight [Mean (Standard Deviation); unit: kg] | 83.2 (14.9) | 77.9 (15.6) | 79.5 (14.5) | 80.5 (15.5) | 78.8 (14.7) | 80.0 (15.1)
Height [Mean (Standard Deviation); unit: cm] | 169.6 (9.5) | 168.2 (9.2) | 167.8 (8.4) | 170.0 (9.8) | 167.9 (9.7) | 168.7 (9.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (4.0) | 27.4 (4.3) | 28.2 (4.3) | 27.8 (4.6) | 27.9 (4.0) | 28.0 (4.3)
Time since first diagnosis of asthma [Median (Full Range); unit: months] | 372.3 [16.2 to 823.1] | 372.8 [26.7 to 758.8] | 373.9 [19.6 to 862.7] | 306.6 [30.8 to 862.5] | 385.0 [17.5 to 833.1] | 363.8 [16.2 to 862.7]
Age at first diagnosis of asthma [Mean (Standard Deviation); unit: years] | 17.4 (18.3) | 17.3 (18.1) | 17.2 (17.7) | 17.4 (18.0) | 16.5 (15.8) | 17.2 (17.6)
Asthma medication category at study entry [Count of Participants; unit: Participants]
  Short-Acting β2-agonist (SABA), (albuterol) | 115 | 115 | 117 | 124 | 121 | 592
  Leukotriene Receptor Antagonist (LTRA) | 24 | 7 | 17 | 18 | 17 | 83
  Theophylline | 0 | 0 | 0 | 0 | 0 | 0
  Inhaled Corticosteroid (ICS) alone | 23 | 26 | 34 | 36 | 28 | 147
  ICS/ Long-Acting β2-agonist (LABA), (free or fixed combination) | 93 | 88 | 86 | 88 | 94 | 449
  ICS/Long-Acting Muscarinic Antagonist (LAMA), (free combination) | 0 | 0 | 0 | 0 | 0 | 0
  ICS/LABA/LAMA | 2 | 2 | 0 | 0 | 1 | 5
  Short-Acting Muscarinic Antagonist (SAMA) | 0 | 0 | 0 | 0 | 1 | 1
  SAMA/SABA | 0 | 0 | 1 | 0 | 0 | 1
ICS dose before study [Count of Participants; unit: Participants]
  Low daily dose | 50 | 50 | 48 | 54 | 51 | 253
  Medium daily dose | 68 | 66 | 72 | 70 | 73 | 349
Smoking habits [Count of Participants; unit: Participants]
  Ex-smoker | 13 | 18 | 18 | 21 | 23 | 93
  Non-smoker | 105 | 98 | 102 | 103 | 101 | 509
Duration of smoking [Mean (Standard Deviation); unit: years] — Population: Explain why number analyzed in row differs from overall.
  This was a trial with asthma patients. Only prior smokers were anlayzed for duration of smoking.
  years
    number analyzed (Participants) | 13 | 18 | 18 | 21 | 23 | 93
    (all) | 10.3 (8.2) | 9.5 (6.1) | 13.7 (9.1) | 10.4 (8.6) | 10.3 (6.7) | 10.8 (7.7)
Number of pack-years [Median (Full Range); unit: pack-years] — Measure Description: A pack-year is a term used to describe the approximate number of cigarettes a person has smoked over time. 1 One pack-year equals 20 manufactured cigarettes smoked per day for one year. Population: Explain why number analyzed in row differs from overall. This was a trial of asthma patients. Pack years are only reported for ex-smokers. For one patients in Arm D, the number of pack years was not reported.
  pack-years
    number analyzed (Participants) | 13 | 18 | 18 | 20 | 23 | 92
    (all) | 2.0 [0.5 to 8.0] | 2.7 [0.3 to 8.5] | 4.0 [0.2 to 10.0] | 3.5 [0.2 to 9.0] | 3.0 [0.1 to 8.5] | 3.0 [0.1 to 10.0]
FEV1 at baseline [Mean (Standard Deviation); unit: litres] — Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath during the first second (FEV1).
  litres | 2.131 (0.500) | 2.128 (0.545) | 2.114 (0.531) | 2.268 (0.603) | 2.130 (0.571) | 2.155 (0.553)
FEV1 (% predicted normal value) at baseline [Mean (Standard Deviation); unit: percent of predicted normal value] | 68.5 (8.4) | 68.3 (7.8) | 68.4 (8.7) | 68.6 (8.0) | 68.8 (8.9) | 68.5 (8.4)
FVC at baseline [Mean (Standard Deviation); unit: litres] — Forced vital capacity (FVC) is the maximal volume of gas that can be exhaled from full inhalation by exhaling as forcefully and rapidly as possible.
  litres | 3.159 (0.971) | 3.164 (0.931) | 3.101 (0.855) | 3.415 (1.020) | 3.197 (0.851) | 3.209 (0.931)
FEV1/FVC at baseline [Mean (Standard Deviation); unit: ratio of the parameters] | 0.696 (0.104) | 0.687 (0.099) | 0.693 (0.098) | 0.677 (0.104) | 0.675 (0.106) | 0.685 (0.102)

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose Morning FEV1 at Week 8 - Change From Baseline
Description: Change from baseline in pre-dose morning FEV1 (average of pre-dose FEV1 measurements) at Week 8.
  Spirometry, used to measure FEV1, was performed according to internationally accepted standards.
  Definitions:
  Baseline=Baseline values for pre-dose FEV1 were the average of measurements taken at V2 (Week 0) at 45 minutes and 15 minutes pre-dose; FEV1=Forced expiratory volume in the 1st second;
Time Frame: Baseline, Week 8
Population: Intention to treat:
  All randomized patients who received at least one dose of the study treatment and with at least one available evaluation of efficacy after baseline (primary or secondary efficacy variables) after the baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Groups:
- Treatment A (CHF 718 pMDI 100 µg TDD): CHF 718 pMDI 100 μg Total Daily Dose (TDD), Dose 1;
  CHF 718 pMDI 50 μg/actuation: 1 inhalation 2 times a day (BID);
- Treatment B (CHF 718 pMDI 400 µg TDD): CHF 718 pMDI 400 μg Total Daily Dose (TDD) 400 μg, Dose 2;
  CHF 718 pMDI 100 μg/actuation: 2 inhalations BID;
- Treatment C (CHF 718 pMDI 800 µg TDD): CHF 718 pMDI Total Daily Dose (TDD) 800 μg, Dose 3;
  CHF 718 pMDI 100 μg/actuation: 4 inhalations BID;
- Treatment D (Placebo): Placebo Control. CHF 718 pMDI matched Placebo: 4 inhalations BID;
- Treatment E (QVAR^®, 320 µg TDD): Beclomethasone dipropionate hydrofluoroalkane (HFA) (QVAR^®), Active Control
  Beclomethasone dipropionate hydrofluoroalkane (HFA), Total Daily Dose (TDD) 320 µg; QVAR® 80 μg/actuation: 2 inhalations BID;
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 117 | 115 | 119 | 123 | 124
Litres | 0.021 [-0.036 to 0.077] | 0.090 [0.033 to 0.147] | 0.070 [0.013 to 0.126] | -0.023 [-0.079 to 0.033] | 0.078 [0.024 to 0.133]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.567, Mixed Models Analysis; Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.052 to 0.140]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = 0.113, 95% CI 2-sided [0.018 to 0.209]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [-0.003 to 0.188]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.090, Mixed Models Analysis; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [-0.011 to 0.150]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.231, Mixed Models Analysis; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [-0.031 to 0.129]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.612, Mixed Models Analysis; Mean Difference (Final Values) = -0.021, 95% CI 2-sided [-0.101 to 0.059]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.023 to 0.180]

2. Secondary Outcome: Pre-dose Morning FEV1 at Week 4 - Change From Baseline
Description: Change from baseline in pre-dose morning FEV1 at Week 4.
  Spirometry, used to measure FEV1, was performed according to internationally accepted standards.
  Definitions:
  Baseline=Baseline values for pre-dose FEV1 were the average of measurements taken at V2 (Week 0) at 45 minutes and 15 minutes pre-dose; FEV1=Forced expiratory volume in the 1st second;
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Groups:
- Treatment A (CHF 718 pMDI 100 µg TDD): CHF 718 pMDI 100 μg Total Daily Dose (TDD), Dose 1;
  CHF 718 pMDI 50 μg/actuation: 1 inhalation twice daily (BID);
- Treatment E (QVAR^®, 320 µg TDD): Beclomethasone dipropionate hydrofluoroalkane (HFA) (QVAR^®), Active Control
  Beclomethasone dipropionate hydrofluoroalkane (HFA), Total Daily Dose (TDD) 320 µg; QVAR^® 80 μg/actuation: 2 inhalations BID;
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 117 | 115 | 119 | 123 | 124
Litres | 0.021 [-0.035 to 0.077] | 0.120 [0.064 to 0.177] | 0.073 [0.018 to 0.129] | 0.003 [-0.052 to 0.058] | 0.077 [0.023 to 0.131]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.647, Mixed Models Analysis; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.060 to 0.097]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [0.039 to 0.196]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.076, Mixed Models Analysis; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.008 to 0.149]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 0.099, 95% CI 2-sided [0.020 to 0.179]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.192, Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.026 to 0.131]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.244, Mixed Models Analysis; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.126 to 0.032]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.060, Mixed Models Analysis; Mean Difference (Final Values) = 0.074, 95% CI 2-sided [-0.003 to 0.151]

3. Secondary Outcome: Pre-dose Morning FVC at Week 4 and 8 - Change From Baseline
Description: Change from baseline in pre-dose morning FVC at Week 4 and 8.
  Spirometry, used to measure FVC, was performed according to internationally accepted standards.
  Definitions:
  Baseline=Baseline values for pre-dose FVC were the average of measurements taken at V2 (Week 0) at 45 minutes and 15 minutes pre-dose; FVC=Forced vital capacity;
Time Frame: Baseline, Week 4, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 117 | 115 | 119 | 123 | 124
Litres
  Week 4 | 0.036 [-0.026 to 0.097] | 0.099 [0.037 to 0.161] | 0.066 [0.006 to 0.127] | 0.023 [-0.037 to 0.084] | 0.056 [-0.004 to 0.115]
  Week 8 | 0.014 [-0.053 to 0.080] | 0.089 [0.022 to 0.156] | 0.036 [-0.030 to 0.103] | -0.016 [-0.082 to 0.050] | 0.063 [-0.001 to 0.127]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Week 4 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.780, Mixed Models Analysis; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.074 to 0.098]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Week 4 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.086, Mixed Models Analysis; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [-0.011 to 0.162]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Week 4 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.324, Mixed Models Analysis; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.043 to 0.129]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Week 4 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.153, Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [-0.024 to 0.150]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 4 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.482, Mixed Models Analysis; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.055 to 0.117]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 4 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.463, Mixed Models Analysis; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.119 to 0.054]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Week 4 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.453, Mixed Models Analysis; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [-0.052 to 0.117]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Week 8 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.533, Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.064 to 0.123]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Week 8 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [0.011 to 0.199]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Week 8 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.274, Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.041 to 0.146]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Week 8 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.119, Mixed Models Analysis; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [-0.019 to 0.169]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 8 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.638, Mixed Models Analysis; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.071 to 0.116]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 8 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.274, Mixed Models Analysis; Mean Difference (Final Values) = -0.052, 95% CI 2-sided [-0.147 to 0.042]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Week 8 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.092, Mixed Models Analysis; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.013 to 0.171]

4. Secondary Outcome: Asthma Control Questionnaire-7© (ACQ-7) Score at Week 4 and Week 8 - Change From Baseline
Description: The ACQ consists of 7 items: 6 simple self-administered questions referring to asthma control and rescue treatment usage with 1 week recall, and a 7th item consisting of the percent (%) predicted FEV1 completed by clinic staff. Scoring uses a 7-point scale: 0 = "totally controlled" and 6 = "severely uncontrolled". The ACQ score was calculated as the average of all 7 items.
  Definitions:
  ACQ-7 score=Asthma Control Questionnaire-7©; Information regarding the American Thoracic Society ACQ questionnaire is also available at: https://member.thoracic.org/members/assemblies/assemblies/srn/questionaires/acq.php; Baseline ACQ-7 score = ACQ score recorded at V2 (Week 0) Day 1, before randomization; FEV1=Forced expiratory volume in the 1st second;
Time Frame: Baseline, Week 4, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 117 | 115 | 119 | 123 | 124
score on a scale
  Week 4 | -0.43 [-0.54 to -0.32] | -0.53 [-0.65 to -0.42] | -0.49 [-0.60 to -0.38] | -0.27 [-0.38 to -0.17] | -0.47 [-0.58 to -0.36]
  Week 8 | -0.53 [-0.65 to -0.42] | -0.58 [-0.70 to -0.46] | -0.66 [-0.78 to -0.55] | -0.43 [-0.54 to -0.31] | -0.64 [-0.75 to -0.53]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Week 4 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.053, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.31 to 0.00]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Week 4 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.42 to -0.11]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Week 4 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.37 to -0.06]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Week 4 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.176, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.26 to 0.05]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 4 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.423, Mixed Models Analysis; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.22 to 0.09]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 4 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.574, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.11 to 0.20]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Week 4 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.35 to -0.05]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Week 8 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo; Test type: Superiority; p = 0.215, Mixed Models Analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.27 to 0.06]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Week 8 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.070, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.32 to 0.01]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Week 8 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.40 to -0.07]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Week 8 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.566, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.21 to 0.12]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 8 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.124, Mixed Models Analysis; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.29 to 0.04]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Week 8 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.336, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.25 to 0.08]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Week 8 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.37 to -0.05]

5. Secondary Outcome: Average Use of Rescue Medication - Change From Baseline
Description: Change from baseline in average use of rescue medication, during Inter-visit period 1, Inter-visit period 2, Entire treatment period.
  Definitions:
  Baseline=For the efficacy variable -- average use of rescue medication -- derived from the electronic diary (eDiary), baseline values were the averages recorded during the run-in period;
  Inter-visit period 1=Starts from the pm assessment of the Start of the Randomized Treatment Period to the am assessment at Visit 3 (Week 4);
  Inter-visit Period 2=Starts from the pm assessment of the day the subject returns to the clinic (Visit 3) to the am assessment of the date of Visit 4 (Week 8);
  Entire treatment period=Average of 8 weeks;
  am=morning pm=evening
Time Frame: Baseline (average of the 2-week run-in period); Inter-visit period 1 (average of the first 4 weeks); Inter-visit period 2 (average of the last 4 weeks); Entire treatment period (average of 8 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: puffs/day
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 118 | 115 | 118 | 124 | 124
puffs/day
  Inter-visit period 1 | -0.11 [-0.25 to 0.03] | -0.27 [-0.41 to -0.12] | -0.14 [-0.28 to 0.00] | 0.07 [-0.07 to 0.21] | -0.13 [-0.26 to 0.01]
  Inter-visit period 2 | -0.12 [-0.29 to 0.05] | -0.35 [-0.52 to -0.18] | -0.25 [-0.42 to -0.08] | 0.01 [-0.15 to 0.18] | -0.18 [-0.34 to -0.01]
  Entire treatment period | -0.11 [-0.26 to 0.03] | -0.31 [-0.46 to -0.16] | -0.20 [-0.34 to -0.05] | 0.04 [-0.10 to 0.19] | -0.15 [-0.29 to -0.01]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.067, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.38 to 0.01]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.53 to -0.14]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.038, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.40 to -0.01]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.130, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.35 to 0.05]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.811, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.22 to 0.17]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.202, Mixed Models Analysis; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.07 to 0.33]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.044, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.39 to -0.01]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.283, Mixed Models Analysis; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.37 to 0.11]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.60 to -0.13]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.027, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.50 to -0.03]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.054, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.48 to 0.00]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.258, Mixed Models Analysis; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.38 to 0.10]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.423, Mixed Models Analysis; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.14 to 0.34]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.111, Mixed Models Analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.42 to 0.04]
Statistical Analysis 15: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Entire treatment period Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.135, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.36 to 0.05]
Statistical Analysis 16: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Entire treatment period Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.56 to -0.14]
Statistical Analysis 17: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Entire treatment period Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.44 to -0.03]
Statistical Analysis 18: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Entire treatment period Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.067, Mixed Models Analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.40 to 0.01]
Statistical Analysis 19: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Entire treatment period Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment A (CHF 718 pMDI 100 µg TDD); Test type: Superiority; p = 0.444, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.29 to 0.13]
Statistical Analysis 20: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); Entire treatment period Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); Test type: Superiority; p = 0.285, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.09 to 0.32]
Statistical Analysis 21: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.060, Mixed Models Analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.40 to 0.01]

6. Secondary Outcome: Percentage (%) of Rescue Medication-free Days - Change From Baseline
Description: Change from baseline in percentage (%) of rescue medication-free days. An increased value indicates improvement from baseline.
  Definitions:
  Baseline=For the efficacy variable -- percentage (%) of rescue medication-free days -- derived from the electronic diary (eDiary), baseline values were the averages/percentages recorded during the run-in period.
  Inter-visit period 1=Starts from the pm assessment of the Start of the Randomized Treatment Period to the am assessment at Visit 3 (Week 4);
  Inter-visit Period 2=Starts from the pm assessment of the day the subject returns to the clinic (Visit 3) to the am assessment of the date of Visit 4 (Week 8);
  Entire treatment period=Average of 8 weeks;
  am=morning pm=evening
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: % of rescue medication-free days
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 118 | 115 | 118 | 124 | 124
% of rescue medication-free days
  Inter-visit period 1 | 5.9 [1.9 to 9.9] | 9.0 [5.0 to 13.0] | 6.1 [2.1 to 10.1] | 1.5 [-2.4 to 5.3] | 7.7 [3.9 to 11.6]
  Inter-visit period 2 | 8.9 [4.5 to 13.3] | 13.1 [8.7 to 17.6] | 10.0 [5.6 to 14.4] | 4.1 [-0.2 to 8.4] | 11.2 [7.0 to 15.5]
  Entire treatment period | 7.4 [3.4 to 11.3] | 11.1 [7.1 to 15.1] | 8.1 [4.1 to 12.0] | 2.8 [-1.1 to 6.6] | 9.5 [5.6 to 13.3]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.115, Mixed Models Analysis; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [-1.1 to 10.0]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [2.0 to 13.1]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.099, Mixed Models Analysis; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-0.9 to 10.2]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.275, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-2.5 to 8.8]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.943, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-5.4 to 5.8]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.308, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-8.6 to 2.7]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.024, Mixed Models Analysis; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [0.8 to 11.7]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.129, Mixed Models Analysis; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-1.4 to 11.0]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 9.0, 95% CI 2-sided [2.8 to 15.2]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-0.3 to 12.1]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = 0.180, Mixed Models Analysis; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-2.0 to 10.5]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = 0.721, Mixed Models Analysis; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-5.1 to 7.4]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.328, Mixed Models Analysis; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-9.4 to 3.1]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [1.0 to 13.2]
Statistical Analysis 15: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 15]; Test type: Superiority; p = 0.101, Mixed Models Analysis; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-0.9 to 10.1]
Statistical Analysis 16: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [2.8 to 13.9]
Statistical Analysis 17: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.061, Mixed Models Analysis; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-0.2 to 10.8]
Statistical Analysis 18: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 18]; Test type: Superiority; p = 0.196, Mixed Models Analysis; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-1.9 to 9.3]
Statistical Analysis 19: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 19]; Test type: Superiority; p = 0.814, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-4.9 to 6.3]
Statistical Analysis 20: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 20]; Test type: Superiority; p = 0.291, Mixed Models Analysis; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-8.6 to 2.6]
Statistical Analysis 21: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = 6.7, 95% CI 2-sided [1.3 to 12.1]

7. Secondary Outcome: Overall Daily Asthma Symptoms Scores - Change From Baseline
Description: Overall daily asthma symptoms scores - Change From Baseline (am and pm).
  Subjects had to record asthma symptom score (overall symptoms, cough, wheeze, chest tightness and breathlessness) in the am (night-time asthma symptom score) and in the pm (daytime asthma symptom score). These data were collected in the subject's diary. Daily asthma symptoms score were performed separately for am score and pm score and also as a total, where the total equals the sum of the am and pm scores. Degree of asthma symptoms by score: 0=None, 1=Mild, 2=Moderate, and 3=Severe.
  Baseline=Averages values during the run-in period;
  Inter-visit period 1=Starts from the pm assessment of the Start of the Randomized Treatment Period to the am assessment at Visit 3 (Week 4);
  Inter-visit Period 2=Starts from the pm assessment of the day the subject returns to the clinic (Visit 3) to the am assessment of the date of Visit 4 (Week 8);
  Entire treatment period=Average of 8 weeks;
  am=morning pm=evening
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 118 | 115 | 118 | 124 | 124
score on a scale
  Inter-visit period 1 | -0.1 [-0.1 to -0.0] | -0.1 [-0.1 to -0.0] | -0.1 [-0.1 to -0.0] | 0.0 [-0.0 to 0.1] | -0.1 [-0.2 to -0.1]
  Inter-visit period 2 | -0.1 [-0.2 to -0.1] | -0.1 [-0.2 to -0.1] | -0.1 [-0.2 to -0.1] | -0.0 [-0.1 to 0.0] | -0.1 [-0.2 to -0.1]
  Entire treatment period | -0.1 [-0.1 to -0.1] | -0.1 [-0.1 to -0.1] | -0.1 [-0.2 to -0.1] | 0.0 [-0.0 to 0.1] | -0.1 [-0.2 to -0.1]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.913, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.871, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.958, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = 0.996, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = 0.632, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.630, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]
Statistical Analysis 15: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 15]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0]
Statistical Analysis 16: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.0]
Statistical Analysis 17: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]
Statistical Analysis 18: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 18]; Test type: Superiority; p = 0.960, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 19: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 19]; Test type: Superiority; p = 0.725, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 20: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 20]; Test type: Superiority; p = 0.764, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 21: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to -0.1]

8. Secondary Outcome: Percentage (%) of Asthma Symptoms-free Days - Change From Baseline
Description: Change from baseline in Percentage (%) of asthma symptoms-free days.
  Asthma symptoms-free days is the number of days with a total asthma score=0 (daily morning plus evening asthma score).
  Subjects recorded asthma symptom score as described in the Outcome measure #7.
  Definitions:
  Baseline=For the efficacy variables -- daytime and night-time asthma symptom scores -- derived from the eDiary, baseline values were the averages/percentages recorded during the run-in period;
  Inter-visit period 1=Starts from the pm assessment of the Start of the Randomized Treatment Period to the am assessment at Visit 3 (Week 4);
  Inter-visit Period 2=Starts from the pm assessment of the day the subject returns to the clinic (Visit 3) to the am assessment of the date of Visit 4 (Week 8);
  Entire treatment period=Average of 8 weeks;
  am=morning pm=evening
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: % of of asthma symptom-free days
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 118 | 115 | 118 | 124 | 124
% of of asthma symptom-free days
  Inter-visit period 1 | 8.6 [4.5 to 12.7] | 10.5 [6.4 to 14.7] | 10.1 [6.0 to 14.2] | 5.7 [1.6 to 9.7] | 12.8 [8.8 to 16.8]
  Inter-visit period 2 | 16.4 [11.1 to 21.7] | 17.0 [11.6 to 22.4] | 17.2 [11.8 to 22.51] | 11.7 [6.5 to 16.9] | 21.2 [16.1 to 26.4]
  Entire treatment period | 12.5 [8.0 to 17.0] | 13.8 [9.3 to 18.3] | 13.6 [9.2 to 18.1] | 8.7 [4.3 to 13.1] | 17.0 [12.7 to 21.4]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.316, Mixed Models Analysis; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-2.8 to 8.7]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [-0.9 to 10.7]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.128, Mixed Models Analysis; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [-1.3 to 10.2]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.511, Mixed Models Analysis; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-3.9 to 7.8]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.610, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-4.3 to 7.3]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.882, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-6.3 to 5.4]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 1 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = 7.2, 95% CI 2-sided [1.5 to 12.9]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.219, Mixed Models Analysis; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-2.8 to 12.2]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.166, Mixed Models Analysis; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-2.2 to 12.8]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.151, Mixed Models Analysis; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-2.0 to 12.9]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = 0.871, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-6.9 to 8.2]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = 0.837, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-6.8 to 8.3]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.966, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-7.4 to 7.7]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = 9.5, 95% CI 2-sided [2.1 to 16.9]
Statistical Analysis 15: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 15]; Test type: Superiority; p = 0.233, Mixed Models Analysis; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-2.5 to 10.1]
Statistical Analysis 16: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.113, Mixed Models Analysis; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [-1.2 to 11.4]
Statistical Analysis 17: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.120, Mixed Models Analysis; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [-1.3 to 11.2]
Statistical Analysis 18: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 18]; Test type: Superiority; p = 0.691, Mixed Models Analysis; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-5.1 to 7.6]
Statistical Analysis 19: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 19]; Test type: Superiority; p = 0.722, Mixed Models Analysis; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-5.2 to 7.5]
Statistical Analysis 20: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 20]; Test type: Superiority; p = 0.966, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-6.5 to 6.2]
Statistical Analysis 21: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [2.2 to 14.5]

9. Secondary Outcome: Percentage (%) of Asthma Control Days - Change From Baseline
Description: Change from baseline in percentage (%) of asthma control days, during Inter-visit period 1, Inter-visit period 2, Entire treatment period.
  This outcome measure was calculated according to the following definition: Days with a total daily morning + evening asthma score = 0 AND No rescue medication use.
  Definitions:
  Baseline=For the efficacy variable -- asthma control days -- derived from the eDiary, baseline values were the averages/percentages recorded during the run-in period;
  Inter-visit period 1=Starts from the pm assessment of the Start of the Randomized Treatment Period to the am assessment at Visit 3 (Week 4);
  Inter-visit Period 2=Starts from the pm assessment of the day the subject returns to the clinic (Visit 3) to the am assessment of the date of Visit 4 (Week 8);
  Entire treatment period=Average of 8 weeks;
  am=morning pm=evening
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: % of asthma control days
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 118 | 115 | 118 | 124 | 124
% of asthma control days
  Inter-visit period 1 | 7.3 [3.3 to 11.3] | 10.6 [6.5 to 14.6] | 10.4 [6.4 to 14.5] | 5.0 [1.1 to 9.0] | 12.8 [8.8 to 16.7]
  Inter-visit period 2 | 14.3 [9.1 to 19.5] | 16.3 [11.0 to 21.5] | 17.5 [12.2 to 22.7] | 10.5 [5.3 to 15.6] | 20.63 [15.6 to 25.7]
  Entire treatment period | 10.8 [6.4 to 15.2] | 13.4 [9.0 to 17.9] | 13.9 [9.5 to 18.3] | 7.7 [3.4 to 12.1] | 16.7 [12.4 to 21.0]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.426, Mixed Models Analysis; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-3.4 to 7.9]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.055, Mixed Models Analysis; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [-0.1 to 11.2]
Statistical Analysis 3: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.059, Mixed Models Analysis; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [-0.2 to 11.1]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.263, Mixed Models Analysis; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-2.5 to 9.0]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.280, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-2.6 to 8.8]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.965, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-5.9 to 5.6]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 1 Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [2.2 to 13.3]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.308, Mixed Models Analysis; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-3.5 to 11.2]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.124, Mixed Models Analysis; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-1.6 to 13.2]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.063, Mixed Models Analysis; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [-0.4 to 14.3]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = 0.602, Mixed Models Analysis; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-5.5 to 9.4]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = 0.402, Mixed Models Analysis; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [-4.3 to 10.6]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.753, Mixed Models Analysis; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-6.3 to 8.6]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 10.2, 95% CI 2-sided [2.9 to 17.4]
Statistical Analysis 15: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 15]; Test type: Superiority; p = 0.331, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-3.1 to 9.2]
Statistical Analysis 16: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.073, Mixed Models Analysis; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-0.5 to 11.9]
Statistical Analysis 17: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.048, Mixed Models Analysis; Mean Difference (Final Values) = 6.2, 95% CI 2-sided [0.1 to 12.4]
Statistical Analysis 18: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 18]; Test type: Superiority; p = 0.410, Mixed Models Analysis; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-3.6 to 8.9]
Statistical Analysis 19: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 19]; Test type: Superiority; p = 0.320, Mixed Models Analysis; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [-3.1 to 9.4]
Statistical Analysis 20: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 20]; Test type: Superiority; p = 0.867, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-5.7 to 6.8]
Statistical Analysis 21: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 9.0, 95% CI 2-sided [2.9 to 15.0]

10. Secondary Outcome: Pre-dose Peak Expiratory Flow (PEF) (L/Min) (Morning and Evening) - Change From Baseline
Description: Change from baseline in pre-dose Peak Expiratory Flow (PEF) (Liters/min), morning and evening measurements.
  Definitions:
  Baseline=For the efficacy variable -- morning and evening PEF -- derived from the eDiary, the baseline values were the averages/percentages recorded during the run-in period; PEF=evening peak expiratory flow;
  Inter-visit period 1=Starts from the pm assessment of the Start of the Randomized Treatment Period to the am assessment at Visit 3 (Week 4);
  Inter-visit Period 2=Starts from the pm assessment of the day the subject returns to the clinic (Visit 3) to the am assessment of the date of Visit 4 (Week 8);
  Entire treatment period=Average of 8 weeks;
  am=morning pm=evening
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/min
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 116 | 114 | 115 | 121 | 119
Liters/min
  Inter-visit period 1 | -2 [-7.1 to 3.7] | -3 [-8.1 to 2.73] | -4 [-9.3 to 1.5] | -6 [-11.3 to -0.8] | 0 [-5.0 to 5.6]
  Inter-visit period 2 | -4 [-10.9 to 2.3] | 3 [-3.3 to 10.0] | -5 [-11.7 to 1.6] | -4 [-10.3 to 2.8] | 2 [-4.2 to 8.8]
  Entire treatment period | -3 [-8.6 to 2.6] | 0.3 [-5.3 to 6.0] | -4 [-10.0 to 1.1] | -4.9 [-10.4 to 0.6] | 1 [-4.2 to 6.8]
Statistical Analysis 1: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.260, Mixed Models Analysis; Mean Difference (Final Values) = 4, 95% CI 2-sided [-3.2 to 11.9]
Statistical Analysis 2: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.387, Mixed Models Analysis; Mean Difference (Final Values) = 3, 95% CI 2-sided [-4.2 to 10.9]
Statistical Analysis 3: Comparison: Treatment D (Placebo); Inter-visit period 1 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.574, Mixed Models Analysis; Mean Difference (Final Values) = 2, 95% CI 2-sided [-5.4 to 9.7]
Statistical Analysis 4: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = 0.799, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-8.6 to 6.7]
Statistical Analysis 5: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.577, Mixed Models Analysis; Mean Difference (Final Values) = -2, 95% CI 2-sided [-9.8 to 5.5]
Statistical Analysis 6: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = 0.764, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-8.8 to 6.5]
Statistical Analysis 7: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 1 Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Final Values) = 6, 95% CI 2-sided [-1.1 to 13.8]
Statistical Analysis 8: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.908, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-9.9 to 8.8]
Statistical Analysis 9: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.135, Mixed Models Analysis; Mean Difference (Final Values) = 7, 95% CI 2-sided [-2.2 to 16.5]
Statistical Analysis 10: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); Inter-visit period 2 Comparison treatment groups were: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo; Test type: Superiority; p = 0.786, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-10.7 to 8.1]
Statistical Analysis 11: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = 0.109, Mixed Models Analysis; Mean Difference (Final Values) = 8, 95% CI 2-sided [-1.7 to 17.1]
Statistical Analysis 12: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = 0.876, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-10.1 to 8.7]
Statistical Analysis 13: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.080, Mixed Models Analysis; Mean Difference (Final Values) = -8, 95% CI 2-sided [-17.9 to 1.0]
Statistical Analysis 14: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Inter-visit period 2 Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.202, Mixed Models Analysis; Mean Difference (Final Values) = 6, 95% CI 2-sided [-3.2 to 15.3]
Statistical Analysis 15: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 15]; Test type: Superiority; p = 0.635, Mixed Models Analysis; Mean Difference (Final Values) = 2, 95% CI 2-sided [-5.9 to 9.7]
Statistical Analysis 16: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 16]; Test type: Superiority; p = 0.191, Mixed Models Analysis; Mean Difference (Final Values) = 5, 95% CI 2-sided [-2.6 to 13.1]
Statistical Analysis 17: Comparison: Treatment C (CHF 718 pMDI 800 µg TDD) vs Treatment D (Placebo); [analysis description as in outcome 5, analysis 17]; Test type: Superiority; p = 0.914, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-7.4 to 8.3]
Statistical Analysis 18: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment B (CHF 718 pMDI 400 µg TDD); [analysis description as in outcome 5, analysis 18]; Test type: Superiority; p = 0.407, Mixed Models Analysis; Mean Difference (Final Values) = 3, 95% CI 2-sided [-4.6 to 11.3]
Statistical Analysis 19: Comparison: Treatment A (CHF 718 pMDI 100 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 19]; Test type: Superiority; p = 0.718, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI 2-sided [-9.4 to 6.4]
Statistical Analysis 20: Comparison: Treatment B (CHF 718 pMDI 400 µg TDD) vs Treatment C (CHF 718 pMDI 800 µg TDD); [analysis description as in outcome 5, analysis 20]; Test type: Superiority; p = 0.235, Mixed Models Analysis; Mean Difference (Final Values) = -5, 95% CI 2-sided [-12.7 to 3.1]
Statistical Analysis 21: Comparison: Treatment D (Placebo) vs Treatment E (QVAR^®, 320 µg TDD); Entire treatment period Comparison treatment groups were: Treatment E (QVAR^®, 320 µg TDD) vs Treatment D (Placebo); Test type: Superiority; p = 0.118, Mixed Models Analysis; Mean Difference (Final Values) = 6, 95% CI 2-sided [-1.6 to 13.9]

11. Secondary Outcome: Vital Signs (Systolic and Diastolic Blood Pressure) - Change From Baseline
Description: Vital signs (systolic and diastolic blood pressure) at baseline, week 4, and week 8.
  Change from baseline.
  Definitions:
  Baseline=Baseline values were defined at visit 2 (Week 0) pre-dose; DBP=Diastolic blood pressure; SBP=Systolic blood pressure;
Time Frame: Baseline, Week 4, Week 8
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 117 | 115 | 119 | 124 | 124
mmHg
  SBP, Week 4 | -0.4 [-39 to 30] | 1.0 [-18 to 27] | 0.5 [-25 to 24] | 0.6 [-24 to 27] | 0.0 [-20 to 30]
  SBP, Week 8: number analyzed (Participants) | 112 | 111 | 112 | 113 | 121
  SBP, Week 8 | 1.0 [-23 to 30] | 2.5 [-24 to 24] | 0.8 [-32 to 33] | 0.2 [-21 to 34] | -0.9 [-23 to 22]
  DBP, Week 4 | -0.1 [-19 to 20] | 0.2 [-16 to 28] | -0.8 [-24 to 17] | 0.1 [-15 to 18] | 0.8 [-16 to 36]
  DBP, Week 8: number analyzed (Participants) | 112 | 111 | 112 | 113 | 121
  DBP, Week 8 | 0.8 [-12 to 27] | 1.0 [-20 to 21] | 0.3 [-21 to 21] | -0.5 [-17 to 20] | 1.2 [-20 to 21]

12. Secondary Outcome: 12-lead ECG Parameters - Heart Rate - Change From Baseline
Description: 12-lead electrocardiogram (12-lead ECG) parameter - heart rate (HR) was measured at baseline (Day 1) and Week 8.
  Change from baseline.
  Definitions:
  Baseline=Baseline values were defined at visit 2 (Week 0) pre-dose;
  bpm=Beats per minute;
Time Frame: Baseline, Week 8
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: bpm
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 116 | 115 | 116 | 121 | 122
bpm | 0.6 [-28 to 24] | 0.2 [-25 to 22] | 0.4 [-27 to 29] | 1.2 [-22 to 39] | -0.4 [-23 to 22]

13. Secondary Outcome: 12-lead ECG Parameters - PR, QRS, QTcF - Change From Baseline.
Description: 12-lead electrocardiogram (12-lead ECG) parameters - PR, QRS, QTcF intervals - were measured at baseline (Day 1) and Week 8.
  Changes from baseline.
  Definitions:
  Baseline=Baseline values were defined at visit 2 (Week 0); QTcF=Fridericia-corrected QT interval; msec=Millisecond;
Time Frame: Baseline, Week 8
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 119 | 120 | 121 | 124 | 124
msec
  PR: number analyzed (Participants) | 116 | 115 | 116 | 121 | 122
  PR | -2.6 [-39 to 34] | 1.5 [-38 to 31] | -1.9 [-32 to 54] | -1.3 [-50 to 28] | 1.0 [-43 to 71]
  QRS: number analyzed (Participants) | 116 | 115 | 116 | 121 | 122
  QRS | 0.1 [-48 to 42] | -1.3 [-38 to 25] | 0.9 [-29 to 26] | -0.5 [-30 to 21] | -0.3 [-48 to 25]
  QTcF: number analyzed (Participants) | 116 | 115 | 116 | 121 | 122
  QTcF | 1.6 [-56 to 65] | 0.7 [-32 to 126] | 0.7 [-37 to 45] | 4.6 [-73 to 105] | 1.2 [-32 to 91]

14. Secondary Outcome: 12-lead ECG Parameters - Prolonged QTcF - Change From Baseline
Description: Number of participants with prolonged QTcF. Change from baseline.
  Baseline=Baseline values were defined at visit 2 (Week 0) pre-dose; QTcF=Fridericia-corrected QT interval;
Time Frame: Baseline, Week 8
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 119 | 120 | 121 | 124 | 124
Participants
  QTcF > 30 msec | 6 | 4 | 4 | 9 | 3
  QTcF > 60 msec | 1 | 1 | 0 | 2 | 1

15. Secondary Outcome: 24-hr Urine Free Cortisol - Change From Baseline
Description: 24-hr Urinary Free Cortisol - Change From Baseline.
  For the evaluation of the 24-hr Urine-Free cortisol excretion, 24-hour urine samples were collected. Urine-free cortisol was measured using liquid chromatography-tandem mass spectrometry (LC-MS/MS).
  Definitions:
  Baseline=Baseline values were defined at visit 2 (Week 0) pre-dose;
Time Frame: Baseline, Week 8
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Median (Full Range); unit: nmol/day
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 99 | 108 | 99 | 103 | 111
nmol/day | -3.60 [-175.8 to 6492.9] | -5.35 [-249.5 to 299.5] | -4.10 [-285.1 to 430.3] | 1.40 [-1319.9 to 459.2] | -3.50 [-692.2 to 145.5]

16. Secondary Outcome: 24-hr Creatinine - Change From Baseline.
Description: 24-hr Creatinine - Change From Baseline.
  For the evaluation of the 24-hr creatinine excretion, 24-hour urine sample were collected. Creatinine was measured using liquid chromatography-tandem mass spectrometry (LC-MS/MS).
  Definitions:
  Baseline=Baseline values were defined at visit 2 (Week 0) pre-dose;
Time Frame: Baseline, Week 8
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Median (Full Range); unit: umol/mol
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
Number analyzed (Participants) | 101 | 110 | 104 | 107 | 111
umol/mol | 0.00 [-0.7 to 0.8] | 0.00 [-0.7 to 0.5] | 0.00 [-0.7 to 0.5] | 0.00 [-0.7 to 0.5] | 0.00 [-1.0 to 0.7]

ADVERSE EVENTS:
Time Frame: From the first intake of study medication (visit 2, Week 0) until study completion (Visit 4, week 8) or discontinuation from the study.
Description: The safety population was used for the evaluation of adverse event (AEs). Safety population=All randomized patients who received at least one dose of study treatment.
  The overall number of randomized participants in the study=610 (Participant Flow). Nevertheless, the Safety population=608 patients; 2 patients (1 in Group A and 1 in Group C) were excluded because they were mistakenly randomized; they failed to meet inclusion criterion #4 and were withdrawn prior to study drug administration.
Groups:
- Treatment D (Placebo): Placebo Control, Placebo; CHF 718 pMDI matched Placebo: 4 inhalations BID;
- Treatment E (QVAR^®, 320 µg TDD): QVAR^®, : Active Control
  Beclomethasone dipropionate hydrofluoroalkane (HFA), Total Daily Dose (TDD) 320 µg;
  QVAR® 80 μg/actuation: 2 inhalations BID;
Arm/Group | Treatment A (CHF 718 pMDI 100 µg TDD) | Treatment B (CHF 718 pMDI 400 µg TDD) | Treatment C (CHF 718 pMDI 800 µg TDD) | Treatment D (Placebo) | Treatment E (QVAR^®, 320 µg TDD)
All-Cause Mortality (participants affected / at risk) | 0/119 | 1/120 | 0/121 | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 1/119 | 2/120 | 2/121 | 1/124 | 0/124
Other Adverse Events (participants affected / at risk) | 18/119 | 8/120 | 25/121 | 28/124 | 21/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (CHF 718 pMDI 100 µg TDD) (N=119) | Treatment B (CHF 718 pMDI 400 µg TDD) (N=120) | Treatment C (CHF 718 pMDI 800 µg TDD) (N=121) | Treatment D (Placebo) (N=124) | Treatment E (QVAR^®, 320 µg TDD) (N=124)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (CHF 718 pMDI 100 µg TDD) (N=119) | Treatment B (CHF 718 pMDI 400 µg TDD) (N=120) | Treatment C (CHF 718 pMDI 800 µg TDD) (N=121) | Treatment D (Placebo) (N=124) | Treatment E (QVAR^®, 320 µg TDD) (N=124)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2) | 3 (3) | 3 (3) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1) | 7 (7) | 6 (6) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 5 (5) | 11 (11) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03084718/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03084718/SAP_001.pdf